CLINICAL TRIAL: NCT05071911
Title: Feasability Study of a New Technique of Axillary Evaluation in Patients With Node Positive Breast Cancer Following Neo-adjuvant Chemotherapy
Brief Title: Targeted Axillary Dissection After Neo-adjuvant Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: TADANAC
Record Dates: First submitted 2021-09-27; First posted 2021-10-08 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — DAT protocol 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: TAD (Targeted Axillary Dissection) — Dual agent SLNB + resection of proven lymph nodes metastasis marked with clip at diagnosis

SUMMARY:
Currently most breast cancer patients with confirmed axillary lymph node metastasis (cN1) at diagnosis are candidates for neoadjuvant chemotherapy (NAC). The increased utilization of NAC can be attributed to practical clinical advantages. The increasing use of NAC has, however, introduced questions regarding appropriate loco-regional management, including the optimal surgical approach to the axillary lymph nodes.

According to current guidelines, patients presenting with cN1 disease and treated with NAC, still undergo axillary lymph node dissection (ALND). In forty percent of these patients, however, the investigators see a nodal complete pathological response (ypN0). In certain subgroups, triple negative breast cancer and Her2 amplified breast cancer, this percentage is even higher. The investigators would like to lessen surgical morbidity by performing a targeted axillary dissection. The investigators place a clip in the biopsy-proven lymph node metastasis at diagnosis. After NAC, the investigators perform a dual agent sentinel node procedure and remove the clipped node during the same surgery. When these lymph nodes are microscopically tumor-free, the investigators can abolish an ALND. Targeted axillary dissection after NAC for cN1 disease seems to have acceptable false negative rates in previous trials. The investigators would like to further define patients where an ALND can be safely omitted.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cT1-3N1M0 breast cancer, histopathologically confirmed.
* Age greater than or equal to 18 years and less than or equal to 85 years.
* Necessity and agreement to neoadjuvant chemotherapy

Exclusion Criteria:

* Previous surgery ipsilateral axillary or radiation ipsilateral axillary / chest.
* Extranodal metastases M1
* cN2-3 status
* Breast cancer with direct invasion of chest wall and / or skin cT4
* Disease progression (clinical /radiological) under neoadjuvant treatment
* Pregnancy
* Presence of a pacemaker in the ipsilateral chest wall

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients with confirmed axillary lymph node metastasis (cN1) at diagnosis are candidates for neoadjuvant chemotherapy (NAC). Patients will be included in this study if they are diagnosed with cT1-3N1M0 breast cancer, histopathologically confirmed.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of new surgical technique TAD using Magseed | 90 minutes
  Succesful retrievement of sentinel node and clipped node

SECONDARY OUTCOMES:
Correlation between ITC/ micrometastasis / macrometastasis in retrieved TAD nodes and number of additional lymph node metastasis in ALND | Two weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium